CLINICAL TRIAL: NCT05460260
Title: GlucoMen Day Cascade CGM 21-Day Study
Brief Title: Glucomen Day Cascade CGM System 21-Day Wear Study
Acronym: GLUCODAY21
Status: Completed | Type: Observational
Sponsor: WaveForm Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-19-0037
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2021-10

CONDITIONS: Efficacy of a 21-Day Wear Period for the Cascade CGM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- GLUCODAY21: Study subjects for 21-day study
  Interventions: Device: Cascade CGM

INTERVENTIONS:
Device: Cascade CGM — 21-days of CGM wear

SUMMARY:
Assessment of 21-day CGM wear period

DETAILED DESCRIPTION:
This single-site study will include 10 subjects who will wear two CGMs for 21 days. On day 1, 5, 10, 15, and 21 subjects will be in-clinic for 12 hrs of testing with YSI blood glucose measurements taken every 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of type 1 or type 2 (on insulin therapy) diabetes mellitus for at least 6 months

  * 18 years of age or older
  * Currently self-monitoring capillary blood glucose (on average at least three times per day or more) or on a CGM for at least three months
  * Be willing to have blood glucose levels manipulated into high and low glucose levels during in clinic days if deemed appropriate per the protocol based on insulin use.
  * Willing to follow all study procedures, including attending all clinic visits during which a venous line will be inserted for blood sampling, wearing CGM sensors for entire study, performing fingertip glucose tests for self-monitoring and calibration, and keeping a diary of activities.
  * Be willing to wear two investigational CGM devices.
  * Sign informed consent form

Exclusion Criteria:

* • Known allergy to medical grade adhesives

  * Magnetic Resonance Imaging (MRI) scheduled during CGM sensor wear period
  * Persons with type 2 diabetes using diet and exercise only for diabetes management
  * Used an investigational drug within 30 days prior to study entry
  * Hematocrit < 32% (obtained during screening)
  * Inadequate veins (in the opinion of the investigator) or known contraindication to placement of a dedicated peripheral line for venous blood withdrawal
  * Symptomatic coronary artery disease with a history of angina, or history of a myocardial infarction or coronary intervention (e.g., percutaneous transluminal coronary angioplasty [PTCA], stent placement), or coronary artery bypass graft (CABG) within the past six months
  * Diagnosis of the following diabetic autonomic neuropathies: orthostatic hypotension, heart rate anomalies, gastroparesis
  * Cerebrovascular incident within the past six months
  * History or presence of eczema, psoriasis, atopic or contact dermatitis
  * Pregnancy at the start of the study.
  * Current use or within one-week exposure to topical medications at the proposed insertion sites
  * Seizure disorder (epilepsy)
  * Malignancy within the past five years, except basal cell or squamous cell skin cancers
  * Major surgical operation within 30 days prior to screening
  * Other medical conditions that would pose safety concerns, interfere with study conduct or seriously compromise study integrity (reason for exclusion will be clearly documented by investigator or designee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with Type I and Type II Diabetes
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
21-Day CGM Functionality The secondary objective is: -To evaluate the uniformity of the performance of the WaveForm GlucoMmen Day Cascade CGM over 21 days. | 21 Days
  To evaluate the feasibility of a 21-day wear CGM system.
  The secondary objective is:
  -To evaluate the uniformity of the performance of the WaveForm GlucoMmen Day Cascade CGM over 21 days.
  To evaluate the feasibility of a 21-day wear CGM system.

SECONDARY OUTCOMES:
Evaluation of Uniformity | From 15 to 21 days
  To evaluate the uniformity of the performance of the WaveForm GlucoMen Day Cascade CGM over 21 days.

CONTACTS AND LOCATIONS:
Locations (2):
- Clinical Hospital "Sveti Duh", Zagreb, Croatia
- Miremo, d.o.o, Novo Mesto, Slovenia